CLINICAL TRIAL: NCT04024774
Title: Diagnostic Research in Patients With Rare Diseases -Solving the Unsolved Rare Diseases
Acronym: AnDDI-Solve-RD
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OLIVIER-FAIVRE H2020 2017
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Rare Diseases
MeSH Terms: conditions — Rare Diseases | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- index cases and their parents
  Interventions: Biological: Biological samples; Genetic: Genetic test

INTERVENTIONS:
Biological: Biological samples — blood samples, urine samples, tissue samples
Genetic: Genetic test — anamnesis and NGS sequencing

SUMMARY:
Most diagnostically unsolved rare disease have a genetic cause. These causes have not been found applying the current methodologies due to technical limitations (e.g. repeat expansions, changes in non-coding (intronic) regions) or, although methodically recorded, their pathophysiological significance but not classified as clinically relevant. A re- and meta-analysis of existing data sets with new algorithms and statistical models as well as the complementation with other omics technologies followed by functional follow-up studies in appropriate disease models (e.g. patient cell lines) allows to elucidate additional causes of diseases and improve the diagnosis of hereditary diseases. In addition to the direct examination of persons affected, the analysis of healthy family members, for example of parents, plays an important role in a so-called trio analysis, especially in the efficient filtering of the extensive data sets for newly created changes, so-called de novo- Variants (new mutations). In the context of the outlined analyzes, new disease genes can be found and validated. The gain of scientific knowledge due to a better understanding of basic cell biological mechanisms can contribute to the development of targeted therapeutic approaches.

In this context, the Solve-RD project has been built and financed by the European Union with the ambitions to solve large numbers of rare disease, for which a molecular cause is not known yet by sophisticated combined omics approaches, and to improve diagnostics of rare disease patients. Solve-RD fully integrates with the newly formed European Reference Networks (ERNs) for rare diseases, and in particular the ERN-RND, -EURO-NMD, -ITHACA, and -GENTURIS. The AnDDI-Rares network is fully affiliated to the ERN ITHACA network and will actively contribute to the project, by the ambition of sharing knowledge about genes, genomic variants and phenotypes.

The project will first reanalyse 18.000 negative exomes from the different ERNs performed in a diagnostic or research context (collection of biomaterial, clinical/phenotypic data plus next-generation sequencing has already been performed, and the patient/family has agreed previously in writing that their sample could be used for research related to their disease, with no study related presence required. The project will also propose new multi-omics analyses with new samples needed in 500 patients and their parents in total, justifying the AnDDI-Solve-RD project.

ELIGIBILITY:
Inclusion Criteria:

* Persons or legal guardian who have given their written informed consent
* Unclear molecular cause of the disease corresponding to the list of diseases selected by the Solve-RD data interpretation force (principal investigator part of the team)
* Suspected genetic cause of the disease with negative exome reanalysis
* Healthy parents available for trio analysis

Exclusion Criteria:

* Person not affiliated to a national health insurance scheme

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rare diseases
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Molecular genetic | Day 1
  Verification of the genetic causes of unclear genetic diseases

SECONDARY OUTCOMES:
Number of diagnoses | Day 1
  Improve number of diagnoses of unclear syndromes
Characterization of gene defects | Day 1
  Further characterization of the identified gene defects
Number of patients receiving appropriate therapy after successful diagnosis | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

IPD SHARING:
Plan to Share IPD: No